CLINICAL TRIAL: NCT06211530
Title: Wireless Disposable SpO2 Sensor Hypoxia Testing
Acronym: SpO2 Dispo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2023-061-MS-GES
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: SpO2; Peripheral Oxygen Saturation Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SpO2 Measurements - All Subjects (Experimental): Participants participating in this study will be connected to sensors. The participants are exposed to a desaturation protocol. The protocol is consistent with the ISO 80601-2-61 pulse oximetry standard.
  Interventions: Device: SpO2 Sensor Testing

INTERVENTIONS:
Device: SpO2 Sensor Testing — Participants participating in this study will be connected sensors.The participants are exposed to a desaturation protocol. The protocol is consistent with the ISO 80601-2-61 pulse oximetry standard.

SUMMARY:
The purpose of the study is to collect SpO2 data with simultaneous transfer standard SpO2 measurements data on human participants.

DETAILED DESCRIPTION:
The primary objective of the study is to collect SpO2 data with simultaneous transfer standard SpO2 measurements data (simulating blood sample Spo2) on adult human subjects. Transfer standard is a validated pulse oximetry equipment with a calibration directly traceable to CO-oximetry. Test method and protocol is developed according to ISO 80601-2-61:2017 annex EE.3 (PROCEDURE for non-invasive laboratory testing on healthy adult volunteers) The safety objective is to collect safety information, including type and number of AEs, SAEs, and device issues.

This is a pre-market, open label, prospective, non-randomized clinical research study conducted at one site in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is adult 18-50 years of age.
2. Biological Male or female of any race
3. Participant is a non-smoker or who has not smoked within 2 days prior.
4. Participant must have the ability to understand and provide written informed consent.
5. Participant is adult must be willing and able to comply with study procedures and duration.

Exclusion Criteria:

1. Participant is considered as being morbidly obese (defined as BMI greater than 39.5)
2. Compromised circulation (i.e., Raynaud's Syndrome), injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the particular sites utilized).
3. Tattoo in the optical path which would limit the ability to test sites needed for the study.
4. Females who are pregnant - confirmed by self-performed and self-reported positive urine pregnancy test performed on the day of the study unless the participant is known to be not of child-bearing potential
5. Participants who have smoked in the last 2 days or participants who have refrained, for at least 48 hours, with COHb levels greater than 3% as assessed per site standard operation procedure.
6. Participants with self-reported respiratory conditions such as: uncontrolled/severe asthma, flu, pneumonia/bronchitis, shortness of breath/respiratory distress, unresolved respiratory or lung surgery, emphysema, COPD, lung disease, and/or recent COVID (last 2 months).
7. Participants with self-reported heart or cardiovascular conditions such as: cardiovascular surgery - except successful minor surgery without clinical symptoms (i.e., PFO, PDA), chest pain (angina), previous heart attack, blocked artery, unexplained shortness of breath, congestive heart failure (CHF), history of stroke, transient ischemic attack, carotid artery disease, myocardial ischemia, myocardial infarction, cardiomyopathy, Cardiovascular implantable active medical device (such as pacemaker or automatic defibrillator), Heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia, and/or High blood pressure: systolic greater than140 mmHg or diastolic greater than 90 mmHg on 3 consecutive readings
8. Participants with self-reported health conditions such as: diabetes, uncontrolled thyroid disease, kidney disease/chronic renal impairment, history of seizures (except childhood febrile seizures), epilepsy, history of unexplained syncope, recent history of frequent migraine headaches, recent symptomatic head injury (within the last 2 months), Cancer requiring chemotherapy, radiation, or currently on treatment, Participants with self-reported known clotting disorders, history of bleeding disorders or personal history of prolonged bleeding from injury, history of blood clots, hemophilia, current use of blood thinner: prescription or daily use of aspirin, and/or Sickle Cell Trait or Disease.

10. Participants with severe contact allergies to standard adhesives, latex, silicone, or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported) 11. Unwillingness or inability to remove colored nail polish or non-clear artificial nails from test digits 12. Surgical hardware in pathway which would limit the ability to test sites needed for the study 13. Other known health condition, should be considered upon disclosure in health assessment form.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, NP, Principal Investigator — Element Materials Technology
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foglia EE, Whyte RK, Chaudhary A, Mott A, Chen J, Propert KJ, Schmidt B. The Effect of Skin Pigmentation on the Accuracy of Pulse Oximetry in Infants with Hypoxemia. J Pediatr. 2017 Mar;182:375-377.e2. doi: 10.1016/j.jpeds.2016.11.043. Epub 2016 Dec 9. PMID 27939107
- [Background] Tin W, Lal M. Principles of pulse oximetry and its clinical application in neonatal medicine. Semin Fetal Neonatal Med. 2015 Jun;20(3):192-7. doi: 10.1016/j.siny.2015.01.006. Epub 2015 Feb 18. PMID 25704605
- [Background] Gehring H, Duembgen L, Peterlein M, Hagelberg S, Dibbelt L. Hemoximetry as the "gold standard"? Error assessment based on differences among identical blood gas analyzer devices of five manufacturers. Anesth Analg. 2007 Dec;105(6 Suppl):S24-S30. doi: 10.1213/01.ane.0000268713.58174.cc. PMID 18048894
- [Background] Batchelder PB, Raley DM. Maximizing the laboratory setting for testing devices and understanding statistical output in pulse oximetry. Anesth Analg. 2007 Dec;105(6 Suppl):S85-S94. doi: 10.1213/01.ane.0000268495.35207.ab. PMID 18048904
- [Background] Fouzas S, Priftis KN, Anthracopoulos MB. Pulse oximetry in pediatric practice. Pediatrics. 2011 Oct;128(4):740-52. doi: 10.1542/peds.2011-0271. Epub 2011 Sep 19. PMID 21930554
- See also: FDA -- U.S. Food and Drug Administration. Pulse Oximeters -- Premarket Notification Submissions [510(k)s] - Guidance for Industry and Food and Drug Administration Staff. March 4, 2013. — https://www.fda.gov/downloads/medicaldevices/deviceregulationandguidance/guidancedocuments/ucm081352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 participants were enrolled; 31 subjects completed all study procedures.
Groups:
- SpO2 Measurements - All Subjects: Participants participating in this study will be connected to eight (8) Portrait Mobile P-SA01PL/P-SP01PL prototype sensors provided by GEHC and two reference monitors, Nellcor N-600X V 1.6.0.0 and a forehead sensor, used as standard operating procedures at the site. Data will be collected using the Portrait Hub patient monitor. The participants are exposed to a desaturation protocol that sequentially decreases the SpO2 in a stepwise fashion. The goal is to achieve six stable oxygenation plateaus between 100 and 70% SpO2, while recording simultaneous SpO2 readings from the prototype and reference devices. The protocol is consistent with the ISO 80601-2-61 pulse oximetry standard.
  SpO2 Sensor Testing: Participants participating in this study will be connected to eight (8) Portrait Mobile P-SA01PL/P-SP01PL prototype sensors provided by GEHC and two reference monitors, Nellcor N-600X V 1.6.0.0 and a forehead sensor, used as standard operating procedures at the site. Data will be collected using the Portrait Hub patient monitor. The participants are exposed to a desaturation protocol that sequentially decreases the SpO2 in a stepwise fashion. The goal is to achieve six stable oxygenation plateaus between 100 and 70% SpO2, while recording simultaneous SpO2 readings from the prototype and reference devices. The protocol is consistent with the ISO 80601-2-61 pulse oximetry standard.
Period: Overall Study
Arm/Group | SpO2 Measurements - All Subjects
Started | 32 (32 subjects were enrolled, 31 subjects were analyzed)
Completed | 31
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | SpO2 Measurements - All Subjects
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.42 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31
Skin Pigment [Number; unit: Participants] — Monk Skin Scale was used to to visually assess skin pigment at the forehead to assure enrolment of skin tone diversity. Higher numbers indicate darker skin tones. Lower numbers indicate lighter skin tones.
  Participants
    Monk 01 (Lightest Skin Tone) | 4
    Monk 02 | 4
    Monk 03 | 1
    Monk 04 | 2
    Monk 05 | 5
    Monk 06 | 2
    Monk 07 | 2
    Monk 08 | 7
    Monk 09 | 2
    Monk 10 (Darkest Skin Tone) | 2

OUTCOME MEASURES:

1. Primary Outcome: Collection of Subject SpO2 Percentage Sensor Data With Transfer Standard Measurements for Validation
Description: The collection of SpO2 percentage sensor data with simultaneous transfer standard SpO2 percentage measurements (simulating blood sample SpO2) from each subject enrolled in the study.
Time Frame: 2 Weeks
Measure: Number; unit: data sets
Groups:
- SpO2 Measurements - All Subjects: Subjects participating in this study will be connected to SpO2 sensors. The participants are exposed to a desaturation protocol. The protocol is consistent with the ISO 80601-2-61 pulse oximetry standard.
Arm/Group | SpO2 Measurements - All Subjects
Number analyzed (Participants) | 31
data sets | 31

2. Other Pre Specified Outcome: Number of Safety Events
Description: The collection of the number of adverse events, serious adverse events, and/or device deficiencies reported on all enrolled subjects in the study.
Time Frame: 2 Weeks
Measure: Number; unit: safety events
Groups:
- SpO2 Measurements - All Subjects: Participants participating in this study will be connected to SpO2 sensors. The participants are exposed to a desaturation protocol. The protocol is consistent with the ISO 80601-2-61 pulse oximetry standard.
Arm/Group | SpO2 Measurements - All Subjects
Number analyzed (Participants) | 31
safety events
  Adverse Event | 1
  Serious Adverse Event | 1

ADVERSE EVENTS:
Time Frame: 2 Weeks
Description: All adverse events (AE), including all serious adverse events (SAE), are required to be collected, investigated, and documented. AEs will be collected from [describe the reporting period, e.g., from the time they enter the scan room to the time they leave the scan room]. All AEs will be followed through to their resolution.
Groups:
- Collection of Adverse Events: Collection of all information, including type and number of AEs, SAEs, and device issues.
Arm/Group | Collection of Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 1/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collection of Adverse Events (N=32)
SAE (Cardiac disorders) | 1 (1) — Cardiac arrithymia assessed during monitoring
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collection of Adverse Events (N=32)
AE (Cardiac disorders) | 1 (1) — Cardiac arrithymia assessed during monitoring

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT06211530/Prot_ICF_000.pdf